CLINICAL TRIAL: NCT05379088
Title: Activity Level Monitoring Study
Acronym: ALMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Charles Emery PhD, Professor and Department Chair, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021B0332
Record Dates: First submitted 2022-04-27; First posted 2022-05-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Morbid Obesity
Keywords: sedentary; activity; morbid obesity; obesity; Actigraph
MeSH Terms: conditions — Obesity; Obesity, Morbid; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Additional Follow-up (Experimental): In addition to receiving an ActiGraph activity monitor, participants will complete weekly phone/zoom calls with research staff for a more in-depth monitoring of their activity level.
  Interventions: Behavioral: Phone/zoom calls
- Activity Level Monitoring (No Intervention): Participants receive an ActiGraph activity monitor to track their activity level over a 6-week period.

INTERVENTIONS:
Behavioral: Phone/zoom calls — Participants will complete weekly follow-up phone/zoom calls with a member of the research team. The phone/zoom calls will typically last 30-60 minutes. Participants will discuss barriers to activity and goals for upcoming weeks.
  Arms: Additional Follow-up

SUMMARY:
The purpose of this study is to 1) evaluate the relationship of physical activity to quality of life and psychological functioning among adults with severe obesity (BMI>40) and 2) evaluate the effects of activity monitoring on changes in physical activity during a 6-week intervention interval.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* BMI greater than or equal to 40
* Sit or lie down greater than or equal to 9 hours per day

Exclusion Criteria:

* Participating in regular exercise (any planned exercise)
* Participating in a formal weight loss or exercise program
* Planning to join a formal weight loss or exercise program in the next 2 months
* Cannot stand up without assistance
* Currently pregnant
* Planning to get pregnant in the next 2 months
* Given birth in past 9 months
* Currently breast feeding
* Weigh over 400 lbs
* Highest level of education is below 8th grade
* PHQ-9 score less than 15
* Visual impairment that impairs ability to read
* Any condition(s) that would make it challenging to follow instructions/directions
* Cognitive disorder (e.g., dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Sedentary time | Change from baseline to 6 weeks
  Participants will wear activity monitors for the duration of the study. Sedentary time is operationalized as any recorded waking time spent sitting or lying down.
Sit to stand transitions | Change from baseline to 6 weeks
  Participants will wear activity monitors for the duration of the study. The monitors will keep track of every time a participant goes from sitting to standing and vice versa.
Self-report physical activity | Change from baseline to 6 weeks
  Participants will complete the Modified International Physical Activity Questionnaire - Short Form
Physical function | Change from baseline to 6 weeks
  Participants will complete a 60-foot walk test and 30-second chair stand test.
Health Related Quality of life | Change from baseline to 6 weeks
  Participants will complete the Medical Outcomes Survey, Short Form-36

SECONDARY OUTCOMES:
Perceived stress | Change from baseline to 6 weeks
  Participants will complete the Perceived Stress Scale
Psychological distress | Change from baseline to 6 weeks
  Participants will complete the Hospital and Anxiety Scale
Insomnia | Change from baseline to 6 weeks
  Participants will complete the Insomnia Severity Index
Sleep quality | Change from baseline to 6 weeks
  Participants will complete the Pittsburgh Sleep Quality Index
Pain perception measure 1 | Change from baseline to 6 weeks
  Participants will complete the McGill Pain Questionnaire
Pain perception measure 2 | Change from baseline to 6 weeks
  Participants will complete the Visual Analog Scale for Pain
Weight Stigma measure 1 | Change from baseline to 6 weeks
  Participants will complete the Stigma Situations Inventory
Weight Stigma measure 2 | Change from baseline to 6 weeks
  Participants will complete the Weight Bias Internalization Scale
Weight Stigma measure 3 | Change from baseline to 6 weeks
  Participants will complete the Body Appreciation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Charles Emery, PhD, Principal Investigator — Cardiopulmonary Behavioral Medicine at OSU
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No